CLINICAL TRIAL: NCT03787225
Title: Investigation of Pharmacokinetic Properties, Safety and Tolerability of Single Subcutaneous Doses of NNC0174-0833 in Male Japanese and Caucasian Subjects Being Normal Weight, Overweight or With Obesity
Brief Title: A Research Study of How NNC0174-0833 Behaves in Japanese and Caucasian Volunteers Who Are Normal Weight, Overweight or With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4483; U1111-1219-7303 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-12-21; First posted 2018-12-26 (Actual); Last update posted 2019-06-24 (Actual); Status verified 2019-06

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to 1 of 6 treatment arms, in 3 receiving active NNC0174-0833 and 3 receiving placebo. For statistical analysis and reporting of results, data from the 3 placebo arms will be pooled.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NNC0174-0833 (0.3 mg) (Experimental): Participants will receive single dose of NNC0174-0833
  Interventions: Drug: NNC0174-0833
- NNC0174-0833 (0.9 mg) (Experimental): Participants will receive single dose of NNC0174-0833
  Interventions: Drug: NNC0174-0833
- NNC0174-0833 (1.8 mg) (Experimental): Participants will receive single dose of NNC0174-0833
  Interventions: Drug: NNC0174-0833
- Placebo (NNC0174-0833) (Placebo Comparator): Participants will receive placebo (NNC0174-0833)
  Interventions: Drug: Placebo (NNC0174-0833)

INTERVENTIONS:
Drug: NNC0174-0833 — Participants will receive dose levels of 0.3, 0.9 or 1.8 mg of NNC0174-0833 subcutaneously. Each participant will receive only one dose.
  Arms: NNC0174-0833 (0.3 mg); NNC0174-0833 (0.9 mg); NNC0174-0833 (1.8 mg)
Drug: Placebo (NNC0174-0833) — Participants will receive NNC0174-0833 matched placebo subcutaneously.
  Arms: Placebo (NNC0174-0833)

SUMMARY:
The aim of this study is to look at how the study medicine behaves in the participant's body and how it is removed from the participant's body. The study compares Japanese and Caucasian people who are normal weight, overweight or with obesity. The participants will either get NNC0174-0833 (a potential new medicine) or placebo (a "dummy" medicine similar to the study medicine but without active ingredients) - which treatment any participant gets is decided by chance. Participants will get 1 injection by a study nurse at the clinic. The injection will be with a needle in a skin fold in the participant's stomach area. The study will last for about 4 months, but duration of participation for any participant will last up to about 2 months. The participants will have 8 clinic visits with the study staff.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18-55 years (both inclusive) at the time of signing informed consent.
* For Japanese subjects, both parents of Japanese descent and both paternal and maternal grandparents of Japanese descent.
* For Caucasian subjects, self-reported European descent or white Latin-American descent.
* Body mass index (BMI) between 20.0 and 39.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.
* Body weight between 60 and 110 kg (both inclusive) at screening

Exclusion Criteria:

* Male subject who is not surgically sterilised (vasectomy) and is sexually active (with female partner[s] of childbearing potential), who is not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their non-pregnant female partner(s) (Pearl Index less than 1%), or intend to donate sperm in the period from screening until 3 months following administration of the investigational medical product.
* Any disorder which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-06-04 (Actual)

PRIMARY OUTCOMES:
AUC0-∞,AM833: the area under the NNC0174-0833 plasma concentration-time curve from time 0 to infinity after single dose | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in h*nmol/L

SECONDARY OUTCOMES:
Cmax,AM833: the maximum concentration of NNC0174-0833 in plasma | From Day 1 (pre-dose) until completion of the post-treatment follow-up visit (Day 36)
  Measured in nmol/L
Number of treatment emergent adverse events (TEAEs) | From time of first dosing (Day 1) until completion of the post-treatment follow-up visit (Day 36)
  Count of events

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisktrials.com
URL: http://novonordisk-trials.com